CLINICAL TRIAL: NCT02152904
Title: Risk Factors of Rebleeding After Peptic Ulcer Bleeding: a Nationwide Cohort Study
Acronym: KPUB
Status: Completed | Type: Observational
Sponsor: Joon Sung Kim (Other)
Responsible Party: Sponsor-Investigator, Joon Sung Kim, Clinical assistant proffessor, Department of Internal medicine, Incheon St. Mary's Hospital, Incheon St.Mary's Hospital
Organization: Incheon St.Mary's Hospital (Other)
Other Study IDs: KPUB
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Peptic Ulcer Bleeding
Keywords: Peptic ulcer bleeding; rebleeding; mortality; nationwide
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Peptic ulcer bleeding patients: Endoscopy

SUMMARY:
The purpose of the investigators study is to investigate the factors associated with rebleeding in patients with peptic ulcer bleeding.

DETAILED DESCRIPTION:
The investigators are performing a nationwide population based cohort study to investigate the factors associated with rebleeding in patients with peptic ulcer bleeding. The results of the investigators study should give us information about patients who are at high risk of rebleeindg and enable us to manage these patients appropriately.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with peptic ulcer bleeding by endoscopy
* Patients who consent to be enrolled in the study

Exclusion Criteria:

* Patients who refuse to be enrolled in the study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visit the hospital with symptoms suggestive of peptic ulcer bleeding such as melena or hematemesis. These patients recieve endoscopy and when they are diagnosed with peptic ulcer bleeding are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 892 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Rebleeding rate of peptic ulcer bleeding | 1 year
  The rebleeding rate of patients diagnosed with peptic ulcer ble4eding

SECONDARY OUTCOMES:
Mortality rates of peptic ulcer bleeding | 30 days
  The 30 day mortality rate of patients diagnosed with peptic ulcer bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Wook Kim, Ph.D., Principal Investigator — Incheon St. Mary's Hospital, The Catholic University of Korea
Locations (1):
- Incheon St. Mary's Hospital, Incheon, South Korea